CLINICAL TRIAL: NCT01676168
Title: To Study Gene Expression of Postburn Hypertrophic Scar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205098RIC
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Cicatrix, Hypertrophic
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hypertrophic scar from post-burn patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypertrophic scar: 1x1cm2 hypertrophic scar of post-burn patients are taked by visiting staff when they accept scar-reconstructive surgery.
- normal skin: When the patient accept skin grafting surgery, visiting staff will take 1x1cm2 normal skin.

SUMMARY:
Aim: To compare the gene expression of postburn hypertrophic scar with normal skin.

DETAILED DESCRIPTION:
Background: Postburn hypertrophic scar (HS) remains a challenging problem. Although varied clinical therapeutic methods have been used, none of them has been widely accepted as a standard care. As hypertrophic scar is hereditary, gene therapy can be a potential tool for scar treatment. To investigate the correlation between the clinical presentation of the hypertrophic scar and its gene expression, we propose an analysis of gene expression in the hypertrophic scar using DNA microarray and Real-Time Quantitative PCR. The study result may form the base of clinical treatment.

Methods and Materials: Thirty scar patients requiring surgical treatment in NTUH burn center will be enrolled into the study. Inclusion criteria: (1) Age between 20 and 80 (2) Patients with postburn hypertrophic scar require surgical treatment.

1. Hypertrophic scar and normal skin collection: Under Clinical Trial Informed Consent of Research Ethic Committee, scar and normal skin specimen of 1x1cm2 each will be collected and transported to tissue bank with a vacuum low temperature container. The specimen will be kept in a -80℃ refrigerator.
2. RNA extraction from skin tissue: The RNA extraction will be performed using kit available in the market. Spectrophotometer and gel electrophoresis will be used to measure the purity and concentration of RNA.
3. Gene expression analysis: DNA microarray and Real-Time Quantitative PCR will be used to analyze RNA expression of hypertrophic scar and normal skin.

Statistics: Student's t-test will be used to compare statistically gene expression between hypertrophic scar and normal skin. P < 0.05 will be considered as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* age20~80, hypertrophic scar patient

Exclusion Criteria:

* no specific limitation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient have hypertrophic scar.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kean Eng Yeong, college, Study Chair — NTUH Burn lab
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan